CLINICAL TRIAL: NCT04098822
Title: A 3 Years Naturalistic Cohort Survey Of Virtue® Male Sling System For Male Stress Urinary Incontinence A Post-marketing and Multicenter Prospective Observational Cohort in Subjects With Male Stress Urinary Incontinence
Brief Title: A 3 Years Naturalistic Cohort Survey Of Virtue® Male Sling System For Male Stress Urinary Incontinence
Status: Recruiting | Type: Observational
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: SU018
Record Dates: First submitted 2019-06-07; First posted 2019-09-23 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Urinary Incontinence, Stress
Keywords: Urinary Incontinence, Stress; Suburethral Slings; Prostatectomy
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Virtue male sling — The Coloplast Virtue® Male Sling is a Class II, implantable, sub-urethral, permanent, non-absorbable support sling indicated for the surgical treatment of male SUI resulting from in-trinsic sphincter deficiency (ISD). The sling is manufactured from polypropylene and is sold for single use only. The device is a quadratic sling and consists of a knitted monofilament polypropylene mesh. The body of the device provides surface area for supporting the bulbous urethra.

SUMMARY:
The purpose of this study is to monitor the use of Virtue® Male Sling in a real world population and collect medical data on effectiveness and to monitor safety of Virtue® at 12 and 36 months post device implantation in men with post-prostatectomy urinary incontinence.

DETAILED DESCRIPTION:
This project will be launched after the first introduction of Virtue® Male Sling in Europe. This study is a multicenter prospective, non-interventional (i.e. naturalistic) post-marketing clinical follow up of men with urinary incontinence implanted with Virtue® Male Sling System by urologists who are experienced in the device. The patient will be followed for 12 months in routine real world clinical practice except for administration of subject questionnaire(s). Routine visits will be performed approximately at baseline (preoperative and implantation period), between 1 and 3 months (immediate post-operative period) and 12 months. Then questionnaires will be mailed annually during 2 additional years.

ELIGIBILITY:
Inclusion Criteria:

* Implanted with the Virtue® Male Sling System

Exclusion Criteria:

* Refuses to be included in the survey or that their medical data will be used for research purposes.
* Indication for the Virtue® Male Sling System implantation is not for the treatment of male urinary incontinence

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient implanted with Virtue® Male Sling System to treat post-prostatectomy urinary incontience
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2017-06-29 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Patient Global Impression of Improvement (PGI-I) | 12 months
  PGI-I is a validated questionnaire that collects the patient's impression of improvement after the surgery. Among this 7-point scale (very much better, much better, a little better, no change, a little worse, much worse and very much worse), we ask the patients to check the one number that best decribes how their urinary tract condition is now, compared with how it's was before the surgery. Patients who score little or much or very much better will be considered a treatment success. We measure the percentage of patient who describe the treatment success
Adverse events | 12 months
  Adverse events are any untoward medical occurrence, unintended disease or injury or any untoward clinical signs in subjects. Adverse events will be categorized according to relatedness to device or procedure, severity, and frequency. At 12-months, we measure the percentage of patients without any device related severe or serious adverse events.

SECONDARY OUTCOMES:
Pad weight testing | Baseline, 8 weeks and 12 months
  Percent change in weight from baseline in 24-hour or 1-hour pad weight test
Uroflowmetry | Baseline, 8 weeks, 12 months
  Uroflowmetry including a measure of voided volume and the peak urine flow rate (Qmax) will be collected up to 12-months. Data will be used to determine the presence of urinary obstruction. If the Qmax is considered normal by the physician after the procedure it is not necessary to collect these data at subsequent follow-up visits.
Post-void residual (PVR) volume | Baseline, 8 weeks, 12 months
  PVR volume will be collected pre-and post implant procedure up to 12-months. If the PVR volume is considered normal by the physician after the procedure it is not necessary to collect these data at subsequent follow-up visits.
Pad Use | Baseline, 8 weeks, 12, 24, 36 months
  The number of pads used per day will be collected. Patients will be considered to be pad free if they report never wearing pads or wear pads just for a sense of security.
International Consultation on Incontinence Questionnaire (ICIQ-UI) | Baseline, 8 weeks, 12, 24, 36 months
  The ICIQ-UI Short Form is a self-administred questionnaire to evaluate the frequency, severity, and impact on quality of life of urinary incontinence. Question 1 asked, "How often do you leak urine?" Subjects were instructed to select among "none" (0), "about once a week or less often" (1), "2 or 3 times a week" (2), "about once a day" (3), "several times a day" (4), and "all the time" (5). Question 2 asked, "How much urine do you usually leak (whether you wear protection or not)?" Patients responded with "none" (0), "a small amount" (2), "a moderate amount" (4) or "a large amount (6). Question 3 asked, "Overall, how much does leaking urine interfere with your everyday life?" Participants chose a number from 0 (not at all) to 10 (a great deal). Questions 1, 2 and 3 are summed to compute the total ICIQ SF score. The total score range is then a minimum of 0 to a maximum of 21. The mean score, absolute and relative change compared to baseline will be measure
Subject global satisfaction questionnaire | 8 weeks, 12, 24, 36 months
  This non-validated questionnaire provides additional information concerning patient satisfaction. The survey consists of two questions: How satisfied are you with your surgery?. Among 5 point-scale (very satisfied, satisfied, not satisfied-not dissatisfied, dissatisfied, very dissatisfied), patient check the one item that best describes the subject satisfaction. We measure the percentage the patients who very satisfied and satisfied. The patient answer the question "Do you recommend this operation to a friend?" by yes or no. We measure the percentage the patients who answer "yes".
Incontinence quality of life questionnaire (I-QoL) | Baseline, 8 weeks, 12, 24, 36 months
  The I-QoL is a validated survey questionnaire with 22 items that are scored on a 5-point Likert scale. The I-QOL and its subscale scores are computed by adding each item's response, subtracting the lowest possible score and dividing that sum by the possible raw score range. The scores are then transformed to have a range from 0 (maximum problem) to 100 (no problem at all). The mean score, absolute and relative change compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: René Yiou, Pr, Principal Investigator — CHU Henri Mondor, Créteil, France
Locations (13):
- France (12):
  - CHU Angers, Angers
  - Jean Minjoz Hospital, Besançon
  - CHU de Caen, Caen
  - Centre Hospitalier Chalon Sur Saône William Morey, Chalon-sur-Saône
  - Groupe Hospitalier Henri Mendor, Créteil
  - Claude Huriez Hospital, Lille
  - Clinique Mutualiste de la Porte de l'Orient, Lorient
  - Edouard Herriot Hospital, Lyon
  - Clinique de l'Esperance, Mougins
  - CHU Carémeau, Nîmes
  - Clinique Urologique Nantes-Atlantis, Saint-Herblain
  - Clinique Paul Picquet, Sens
- Ospedale Generale Regionale F. Miull, Acquaviva delle Fonti, Italy

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available